CLINICAL TRIAL: NCT04004104
Title: Design and Rationale for a Randomized Controlled Crossover Trial of Supine Versus Upright Exercise in Patients With Hepatopulmonary Syndrome and Orthodeoxia
Brief Title: Supine Exercise in Hepatopulmonary Syndrome Patients With Orthodeoxia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19-127
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Hepatopulmonary Syndrome
Keywords: Supine Exercise; Orthodeoxia
MeSH Terms: conditions — Hepatopulmonary Syndrome; Platypnea Orthodeoxia Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomized (through a random-number generator, and with cancelled allocation) to start with either an upright exercise test (control arm) or a supine exercise test (intervention arm) on a bicycle ergometer, and then complete the alternate test within 4 weeks.
Who Masked: Outcomes Assessor
Masking Description: The assessor (different from the PI) will not be present when the two exercise tests are performed. Additionally, the results will not be labeled with the specific position of the exercise test. In this manner, the assessor will be blinded to the exercise position and this blinding will strengthen the validity of the research outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control - Upright Exercise (Active Comparator): Participants will perform upright exercise on a cycle ergometer. The opposite test will be completed within 4 weeks.
  Interventions: Diagnostic Test: Upright Exercise
- Intervention - Supine Exercise (Experimental): Participants will perform supine exercise on a cycle ergometer. The opposite test will be completed within 4 weeks.
  Interventions: Diagnostic Test: Supine Exercise

INTERVENTIONS:
Diagnostic Test: Upright Exercise — Exercise is generally performed in the upright position.
  Arms: Control - Upright Exercise
Diagnostic Test: Supine Exercise — Since HPS patients with orthodeoxia experience an improvement in their symptoms and oxygen levels when supine, the intervention will involve them performing exercise in the supine position.
  Arms: Intervention - Supine Exercise

SUMMARY:
Hepatopulmonary syndrome (HPS) is a rare condition that presents in about a quarter of patients with liver cirrhosis. In addition, a small subset of these HPS patients also have orthodeoxia, defined as a drop in oxygen levels when they are sitting up (upright), as opposed to lying flat (supine). At present, there is little known about this condition. Patients diagnosed with HPS and orthodeoxia experience reduced ability to exercise, especially when upright. While standard cardiopulmonary exercise is routinely performed in the sitting position, there are machines that enable candidates to exercise in the supine position. This is especially relevant in patients with severe HPS, with clinically significant orthodeoxia, where conventional upright exercise is difficult. Currently there is a gap in the literature regarding the efficacy of supine exercise compared to upright exercise in these patients. Due to their improvement in dyspnea when lying supine, it is predicted that these patients will be able to exercise for a greater length of time and have increased exercise capacity, which can be projected to improve outcomes pre- and post-transplant.

Overall, HPS patients tend to experience hypoxemia and exercise limitation. Exercise limitation impacts quality of life, incidence and severity of comorbid conditions, and in those who are liver transplant candidates, low exercise tolerance deleteriously impacts transplant outcomes. Accordingly, a strategy that enables patients to exercise more often and/or for longer periods would offer direct benefits to patients with HPS, and if employed as part of an exercise program, could also improve exercise capacity, and thus, liver transplant outcomes.

The purpose of this study is to investigate the effect of supine, compared to upright position on exercise in patients with HPS and orthodeoxia. We hypothesize that these patients will be able to exercise for longer in the supine compared to the upright position, given improved oxygen levels when supine.

DETAILED DESCRIPTION:
This is a 1 year randomized crossover controlled trial study of the effect of supine exercise position (intervention arm) compared to the upright exercise position (control arm) within 4 weeks. This is a single-center study conducted at St. Michael's Hospital, Toronto, Ontario.

The exercise will be performed at a constant work rate, individualized for each participant. Peak work rate will be calculated using results from the most recent room air 6-minute walk test (6MWT), within the past 6 months. The equation used to estimate peak work rate is: Peak Work Rate = 0.168 x 6MWD (m) - 4.085 (ref Kozu Respirology 2010). The individualized constant work rate will be set at 70-80% of this estimated peak work rate.

The main stopping criterion will be the point at which, after standardized encouragement, the subject is unable to continue because of symptoms (i.e. patient does not wish to continue or cannot maintain a minimum peddling frequency of 40 rpm for ≥ 10 seconds). This is defined as the "tolerable limit" (tLIM). Additional safety-related stopping criteria will include: the appearance of life-threatening arrhythmias, a drop in systolic blood pressure by ≥ 10 mm Hg from baseline, or a desaturation below a set point for ≥ 30 s. The set saturation point will be chosen individually for each patient, as the lower of: 80% or the lowest saturation seen on room air 6MWT.

Exercise tests in each position, for each subject, will be standardized with respect to the proper seat adjustment relative to leg length and pedaling cadence (50-60 rpm). Inspiratory capacity will be measured before and after the exercise maneuver.

The cycle ergometer resistance will be set to the pre-determined constant work rate, as described above. There will be continuous monitoring of saturation, ECG, gas exchange, blood pressure, and subjective dyspnea/leg fatigue (Borg scale), with standardized verbal encouragement throughout. Participants will be asked to bring running shoes and comfortable exercise clothes, ensure that they have eaten before the test, to take all usual medications, and to avoid major exercise for 24 hours before the test.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of moderate HPS (defined by liver disease, hypoxemia [PaO2 < 80 mmHg and AaDo2 (alveolar-arterial PO2 difference) ≥ 15 mmHg or ≥ 20 mmHg if age > 64 years] and IPVD (intrapulmonary vasodilatations) as shown by contrast echocardiography])
2. Presence of orthodeoxia (PaO2 decrease by >4 mmHg when patient moves from supine to upright position).

Exclusion Criteria:

1. Pulmonary hypertension (echocardiographic estimated right ventricular systolic pressure >/=50 mmHg and/or right heart catheterization mean pulmonary artery pressure >25 mmHg with pulmonary capillary wedge pressure </= 15 mmHg);
2. Significant obstructive ventilatory impairment (FEV1/FVC ratio < 0.65) (FEV=forced expiratory volume in 1 second; FVC=forced vital capacity)
3. Known significant coronary artery disease;
4. Significant neurologic, orthopedic or rheumatological disorders preventing the use of a cycle ergometer;
5. Other absolute contraindications to submaximal tests (uncontrolled cardiac arrhythmia with hemodynamic compromise, symptomatic severe aortic stenosis, decompensated heart failure and acute cardiopulmonary illness);
6. Moderate or severe ascites.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-07-24 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Stopping time (tLIM) | 12 months
  The main stopping criterion will be the point at which, after standardized encouragement, the subject is unable to continue because of symptoms [defined as the "tolerable limit" (tLIM)]. Additional safety-related stopping criteria will include: the appearance of complex ventricular arrhythmias, intraventricular and/or atrioventricular conduction disorders, bradyarrhythmias, or a desaturation below a set point for ≥ 10 s. The set saturation point will be chosen individually for each patient, as the lower of: 80%, or the nadir desaturation seen on room air six-minute walk test (6MWT).

SECONDARY OUTCOMES:
Isotime Oxygen Uptake (VO2) | 12 months
  Comparing oxygen uptake in the supine and upright position.
Dyspnea | 12 months
  Patient's subjective measure of shortness of breath using Borg scale. This scale ranges from 0 to 10, with 0 being no shortness of breath to 10 being maximal shortness of breath.
Leg Fatigue | 12 months
  Patient's subjective measure of leg fatigue using Borg scale. This scale ranges from 0 to 10, with 0 being no leg fatigue at all to 10 being maximal leg fatigue.
Work Rate | 12 months
  Constant work rate / resistance at which the cycle ergometer was set.
Arterial Oxygen Saturation | 12 months
  The saturation of oxygen in the arteries.
Change in Inspiratory Capacity | 12 months
  Measuring volume of air that can be maximally inspired after normal tidal breaths and comparing between supine and upright.
Reason for Stopping Exercise | 12 months
  Reason due to which tLIM was reached and exercise was stopped.
Minute Ventilation (VE) | 12 months
  The quantity of air expired out of the lungs per minute.
Heart Rate | 12 months
  The number of heart beats per minute, also known as pulse.
VCO2 | 12 months
  Carbon dioxide output per unit of time.
VCO2 over VO2 | 12 months
  The volume of carbon dioxide produced to the volume of oxygen consumed in respiration over a period of time, also known as respiratory quotient (RQ).
HR over VO2 | 12 months
  The change of heart rate to the volume of oxygen consumed in respiration over a period of time.
VE over time | 12 months
  The change of VE during the entire duration of the exercise.
VO2/ HR over time | 12 months
  The change of oxygen pulse during the entire duration of the exercise.
Heart rate over time | 12 months
  The change of heart rate during the entire duration of the exercise.
Cardiac output | 12 months
  The volume of the blood pumped by the heart through the circulatory system in a minute.
Change in inspiratory capacity | 12 months
  The difference of the maximum volume of air that can be inspired following a normal, quiet expiration
VE max | 12 months
  Maximum minute ventilation
End tidal CO2 over time | 12 months
  The point at the end of exhalation when the CO2 reaches its highest concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Samir Gupta, MD, MSc, Principal Investigator — Clinician-Scientist
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parikh H, Lui E, Faughnan ME, Al-Hesayen A, Segovia S, Gupta S. Supine vs upright exercise in patients with hepatopulmonary syndrome and orthodeoxia: study protocol for a randomized controlled crossover trial. Trials. 2021 Oct 9;22(1):683. doi: 10.1186/s13063-021-05633-7. PMID 34625098
- See also: Peak work rate estimated from 6-minute walk distance. — http://www.ncbi.nlm.nih.gov/pubmed/20409022